CLINICAL TRIAL: NCT06381817
Title: Haploidentical Hematopoietic Cell Transplantation Combined With an Unrelated Cord Blood Unit for Acute T Cell Lymphoblastic Leukemia Compared to Haploidentical Hematopoietic Cell Transplantation: a Multicenter, Randomized, Open-label Trial
Brief Title: Haplo-cord HCT vs. Haplo-HCT for T-ALL Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Children's Hospital of Soochow University (Other); Ruijin Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Fujian Medical University Union Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024112
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Acute T Cell Lymphoblastic Leukemia; Haploidentical Hematopoietic Stem Cell Transplantation; Cord Blood
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo-cord HCT (Experimental): Patients enrolled in this arm will receive a coinfusion of cord blood unit in addition to a typical haploidentical hematopoietic cell transplantation
  Interventions: Biological: Haplo-cord HCT
- Haplo-HCT (Active Comparator): Patients enrolled in this arm will receive a typical haploidentical hematopoietic cell transplantation
  Interventions: Biological: Haplo-HCT

INTERVENTIONS:
Biological: Haplo-cord HCT — Haploidentical hematopoietic cell transplantation will be performed with coinfusion of an unrelated cord blood unit
  Arms: Haplo-cord HCT
Biological: Haplo-HCT — Hematopoietic cell transplantation will be performed with a haploidentical donor
  Arms: Haplo-HCT

SUMMARY:
The goal of this clinical trial is to learn if haploidentical hematopoietic cell transplantation combined with an unrelated cord blood unit (haplo-cord HCT) works to treat acute T cell lymphoblastic leukemia (T-ALL). It will also learn about the safety of the transplantation. The main questions it aims to answer are:

Dose co-infusion of cord blood in haploidentical hematopoietic cell transplantation (haplo-HCT) lower the rate of relapse? What medical problems do participants have when having haplo-cord HCT? Researchers will compare haplo-cord HCT to haplo-HCT to see if haplo-cord HCT works to treat T-ALL.

Participants will be infused an unrelated cord blood unit at the same day of haploidentical graft infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute T cell lymphoblastic leukemia
* With available minimal residual disease parameters assessed by flow cytometry and/or quantitative polymerase chain reaction
* Willing to undergo haploidentical hematopoietic cell transplantation and having a suitable haploidentical donor
* With Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Signing an informed consent form, having the ability to comply with study and follow-up procedures

Exclusion Criteria:

* With other malignancies
* Failing to acquire a suitable unrelated cord blood unit
* With a previous history of autologous hematopoietic cell transplantation, allogeneic hematopoietic cell transplantation or chimeric antigen receptor T cell therapy
* With uncontrolled infection intolerant to haploidentical hematopoietic cell transplantation
* With severe organ dysfunction
* In pregnancy or lactation period
* With any conditions not suitable for the trial (investigators' decision)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years after randomization
  estimated progression-free survival at 2 year

SECONDARY OUTCOMES:
Overall survival | 2 years after randomization
  estimated overall survival at 2 year
Cumulative incidence of relapse | 2 years after randomization
  estimated cumulative incidence of relapse at 2 year
Non-relapse mortality | 2 years after randomization
  estimated non-relapse mortality at 2 year
Adverse events | 2 years after randomization
  Number of participants with adverse events. Frequencies of toxicities based on Common Terminology Criteria for Adverse Events (CTCAE) will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Yang XU, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China